CLINICAL TRIAL: NCT05046405
Title: Home-based Transcranial Direct Current Stimulation in Postpartum Depression: the Feasibility Study and Pilot Study
Acronym: 4MUMs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ana Ganho Ávila (Other)
Collaborators: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Sponsor-Investigator, Ana Ganho Ávila, Researcher, University of Coimbra
Organization: University of Coimbra (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020.02059.CEECIND; PTDC/PSI-GER/3110/2021 (Other: Foundation for Science and Technology)
Record Dates: First submitted 2021-07-20; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Postnatal Depression
Keywords: Depression; Postnatal; Postnatal Depression; Transcranial Direct Current Stimulation; Feasibility study; Pilot Study
MeSH Terms: conditions — Depression, Postpartum; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Feasibility studies aim to inform large RCT studies. Thus, for the feasibility study, the investigators aim to inform the practicality of the future Phase-III RCT and to unveil threats to the validity of the efficacy outcomes. Within a users'-centred approach and co-designed methodology, the investigators will assess safety, feasibility of the intervention, and feasibility of procedures for outcomes' assessment. Additionally, the investigators will estimate recruitment/retention and sample size. A consequent underpowered pilot study will be conducted following the achieved static protocol, based on the assumption that the procedures are well defined, serving the purpose of gathering preliminary information and testing the study protocol. Both the feasibility and the pilot studies will be open-label, single arm, single-site longitudinal studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- home-based remotely supervised tDCS (Experimental): The intervention combines home-based tDCS (1 or 2 cycles of 15 daily sessions for 3 weeks/cycle at 2 mA for 30 minutes) with tele-health for remote supervision and e-health for self-monitoring of depressive symptoms.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation (tDCS) has been suggested to the peripartum period combining antidepressant eﬀects with low risks. In tDCS a low intensity constant current is delivered to the scalp with sub-threshold eﬀect on neurons' resting membrane potential. Long stimulation sessions lead to lasting eﬀects and neuroplastic changes. Local tDCS eﬀects target calcium-dependent synaptic plasticity and distal eﬀects alter the networks' connectivity, synchronicity and oscillatory patterns. tDCS applications aim to counteract the hypoactivity of the frontoparietal network and the left sided hyperactivity of the default mode network associated with depressive symptoms.

SUMMARY:
Postpartum Depression (PPD) is a Major Depressive (MD) Disorder occurring within the 12 months after delivery with negative effects to the mother, the child and the family and an estimated prevalence in Europe of 10-15%. Non-invasive Transcranial Direct Current Stimulation (tDCS) has been suggested to PPD, as it combines antidepressant effects with low risks, being equivalent to pharmacotherapy, and showing faster response than psychotherapy. tDCS uses a weak electric current applied to the scalp, modulating neurons' firing rate and neuroplasticity of cerebral circuits to counteract dysfunctional connectivity and inter-hemispheric imbalance in MD. tDCS portability led to its introduction as a home-based intervention and trials assessing home-based tDCS in MD were successful, proved its feasibility and showed good acceptance and benign effect in patients' self-efficacy. Hence, combining home-based tDCS with eHealth systems to support data collection and teleHealth for remote health care has shown positive results in other neuropsychiatric disorders.

To uptake tDCS to PPD, further research is needed. To pursue the needed regulatory steps, current consensus on the primary hypothesis of efficacy is that future phase-III studies must be supported by the identification of biotypes of depression and should include cost-effectiveness analysis to model its economic advantage and inform Health Technology Analysis.

4MUMs, within an iterative user-centred and co-design approach will adopt a combined intervention (home-based tDCS + eHealth system + teleHealth system) for PPD, conduct a dynamic feasibility study of the data collection procedures and intervention, and test these in a single-arm pilot study towards the first large-sample multicentre Phase-III RCT protocol aimed at testing home-based tDCS efficacy in PPD.

DETAILED DESCRIPTION:
Study aims and endpoints:

Aim 1: Conduct a feasibility study to

1. Determine the feasibility and acceptability of the combined intervention in PPD, by estimating the feasibility and acceptability of i) the home-based tDCS intervention; ii) the eHealth system; iii) the teleHealth system, by women and HP.
2. Determine the feasibility and acceptability of data collection and data analysis procedures of outcome and moderator variables for efficacy studies, namely of psychological functioning of mothers and babies (including neurodevelopment), the dyad, cost-benefit, and neuroinflammatory and stress levels; specifically, acceptability and compliance with the procedures will be evaluated
3. Evaluate the safety of the combined intervention in PPD
4. Estimate the parameters for the protocol of the future multicentric RCT aimed to establish the efficacy of the combined intervention

Aim 2: Conduct a pilot study to

a) Gather preliminary evidence of the efficacy of the combined intervention in PPD as measured by psychological functioning of mothers, babies and the dyad, neuroinflammatory and stress levels and quality of life (QoL), and the role of study moderators (genetic/epigenetic profiles of mothers and babies) in affecting main outcomes.

Study design. Feasibility studies aim to inform large RCT studies. Thus, for the feasibility study, the investigators aim to inform the practicality of the future Phase-III RCT and to unveil threats to the validity of the efficacy outcomes. Within a users'-centred approach and co-designed methodology, the investigators will assess safety, feasibility of the intervention, and feasibility of procedures for outcomes' assessment. Additionally, the investigators will estimate recruitment/retention and sample size. A consequent underpowered pilot study will be conducted following the achieved static protocol, based on the assumption that the procedures are well defined, serving the purpose of gathering preliminary information and testing the study protocol. Both the feasibility and the pilot studies will be open-label, single arm, single-site longitudinal studies.

Procedure. 4MUMS is divided in 3 stages:

Month 1-6 - Pre-feasibility study (Tasks 1-5) - 10 stakeholders (3 practitioners, 2 external expert researchers, 2 patients' representatives, 2 woman woman diagnosed with PPD will be recruited to support the identification of the steps, challenges and solutions to adapt a combined procedure to PPD in a co-design approach exploring their views/experiences with the training materials, assessment procedures and the combined intervention (tDCS + ehealth + teleHealth) using Soterix "1X1 tDCS miniCT" device, model 1601 and ELECTRA-RX (Soterix Medical Inc., NY, US).

Month 7-17 - Feasibility study (Tasks 6-12) Up to 15 medication-free women with mild-severe PPD, their babies and their perinatal Health Practitioner (HP) will be recruited. Recruitment will depend on referrals from Ob-Gyn physicians from the DGONR-CHUC. Women will be informed about 4MUMs and, after consenting, will be assessed for eligibility. Eligible women will be invited to participate and complete monthly screening assessments between the third trimester of pregnancy and up to six months after delivery using the Edinburgh Postnatal Depression Scale. When positive (EPDS>10) during pregnancy, women will be asked to go on completing screening across trimesters and will be referred to their perinatal mental health (PMH) team. After delivery, these women may be included in the intervention group (IG) if EPDS>10. Women screening positive in the postpartum will be invited to enter the IG. The HP will be asked to complete acceptability questionnaires at start of the intervention and end of treatment (N=25).

tDCS protocol. tDCS electrodes will be positioned over the dorsolateral prefrontal cortexes (DLPFC), using the Omni-Lateral-Electrode system. OLE results from studies on tDCS montages in the frontal cortex, concluding that current intensity at the DLPFC can be shaped but not focused, balancing increased focality, reduced electric field variability and clinical ease-of-use. The tDCS protocol was selected from previous literature for non-resistant MD and home-based tDCS for MD and will include daily stimulation sessions (2mA, 30 minutes, across three consecutive weeks (5/week). A second tDCS cycle may be repeated if a pre-set benchmark of ≥25% improvement of PPD symptoms is not met at the end of the first cycle.

The tDCS device and the ehealth/teleHealth systems (ELECTRA-RX) are introduced to patients during at-home training. Educational materials are provided through eHealth. tDCS is self-delivered with teleHealth support ensured across the tDCS course. Both eHealth and teleHealth will be delivered through women' cell-phone connected to ELECTRA-RX.

Month 18-34 - Pilot study (Tasks 13-19). Up to 32 medication-free women with mild-severe PPD, their babies and their HP will be recruited. Recruitment, outcomes' assessment procedures and intervention will follow stage 2 adjusted protocol.

Outcomes. Feasibility outcomes will include measures of compliance, acceptability and tolerability for home-based tDCS and for assessment procedures. The multimodal approach to measure the effect of the intervention includes clinical measures of psychological functioning, mother-baby bonding, mothers' levels of neuroinflammatory and stress/cortisol, quality of life (QoL), and child neurodevelopment and temperament. The investigators will study genetic polymorphisms and epigenetic modifications of mothers as moderators of treatment response. The study of child neuroinflammatory, stress/cortisol and epigenetic profiles will support the test of the association between neurodevelopment and mothers' clinical status.

Data analysis. 4MUMs will conduct descriptive analysis for feasibility, estimates of recruitment and retention rates. To observe intervention impact, underpowered analysis will be conducted using repeated measures ANOVA tests (T1,T2/T3/FU) for clinical symptoms, bonding, QoL, stress and neuroinflammatory levels, adjusting to covariates.

Sample size. The sample size for feasibility studies should support the estimate of critical parameters to the necessary degree of precision. For the feasibility study, the investigators will recruit up to 15 participants, until reaching the definite procedures to be tested. The sample size estimate for the pilot study is based on pervious literature, considers just the primary hypothesis of efficacy and accounts for a dropout rate of 20%. The investigators estimate 32 women, to detect an effect size of .60, with a significance alpha level of .05 and .85 power, using repeated measures ANOVA tests. In Coimbra, there are approximately 5000 births per year, which according to the lowest incidence rates in Europe, represent 450 women diagnosed with PPD, around 20% of which with previous psychiatric conditions. However, women naturally hesitate novel treatments, hence the investigators estimate an acceptance rate of 50%, leading to 180 participants/year to be contacted.

Expected results. Our results will inform the multicentred Phase-III RCT protocol in what concerns safety of the procedure, feasibility of the intervention and feasibility of the multimodal approach to measure the impact of tDCS and its moderators. Previous experience suggests that the intervention will be well accepted and tolerated, offering the first step for the development of a novel medication-free intervention, improving the quality of health services while lowering the costs for mothers, families and the health system.

ELIGIBILITY:
Inclusion Criteria:

* Medication-free women with moderate to severe MD episode according to the Montgomery Asberg Depression Rating Scale (MADRS>7), and peripartum onset, diagnosed before delivery or between the second week and month 6 postpartum
* Between 18-45 years of age
* Pregnancy to term
* Uncomplicated delivery to a healthy newborn
* Must be able to manage the technical aspects of the intervention.

Exclusion Criteria:

* tDCS contraindications
* Previous experience with tDCS
* Mental health disorder other than unipolar depression or anxiety
* Suicidal ideation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-02 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention - Number of completed tDCS applications | At end of treatment (cycle 1 or 2; each cycle is 3 weeks)
  Study reports on the number of completed tDCS applications
Change from Baseline on the feasibility of the intervention according to patients. | At baseline, at end of treatment (cycle 1 or 2; each cycle is 3 weeks) and 1 month follow-up.
  The Acceptability Scale for tDCS treatments - patients version (ACCEPT-tDCS) is a 15-item self-report questionnaire on acceptability of tDCS by patients with a minimum score of 15 and a maximum score of 60. Higher scores correspond to increased acceptability.
Change across treatment and follow-up time points on the feasibility of the intervention - Compliance with symptom monitoring | Weekly from week 1 to week 3 (or week 6 if 2 cycles; each cycle is 3 weeks) and at 1 month follow-up
  Study reports on patients compliance with symptom monitoring
Change across treatment and follow-up time points on the feasibility of the assessment procedures - Compliance with outcomes assessment visits | At the end of treatment cycle 1 and the end of treatment cycle 2 (if 2 cycles are prescribed; each cycle is 3 weeks), and at 1 month follow-up
  Study Reports on patients compliance with outcomes assessment visits.
Change from baseline depressive symptoms. | At baseline and weekly, from week 1 to week 3 (or from week 1 to week 6 if 2 cycles were prescribed) and 1 month follow-up
  Change across treatment and follow-up time points on the Edinburgh Postpartum Depression Scale (EPDS), a 10-item questionnaire to assess the presence and severity of clinically relevant depressive symptoms in the prior week using a 4-point scale. Self-report questionnaire to assess depressive symptoms in the postpartum (through e-health). Scores range between 10 and 40 and higher scores correspond to increased presence/severity of depressive symptoms.

SECONDARY OUTCOMES:
Change from Baseline on the feasibility of the intervention according to Health Providers | At baseline, at end of treatment (cycle 1 or 2; each cycle is 3 weeks) and 1 month follow-up.
  The Acceptability Scale for tDCS treatments - Halth Professionals version (ACCEPTpro-tDCS) a 15-item self-report questionnaire on acceptability of tDCS by health professionals with a minimum score of 15 and a maximum score of 60. Higher scores correspond to increased acceptability.
Feasibility of the intervention - tDCS Adverse Effects | Daily during intervention (3 weeks or 6 weeks when adequate) and 1 month follow-up
  tDCS Adverse Effects Questionnaire is a 15-item questionnaire to assess adverse effects of tDCS. Scores range between 0-75, and higher scores correspond to increased adverse effects
Feasibility of the intervention -Health Technology Users' Satisfaction Survey | At the end of treatment (cycle 1 or 2; each cycle is 3 weeks) and 1 month follow-up.
  The survey satisfaction is a 8-item questionnaire on user's satisfaction concerning the combined intervention ranging between 0 and 40, and higher scores correspond to increased satisfaction.
Change from Baseline on the feasibility of the assessment procedures - Acceptability of outcomes assessment visits by women | At baseline, at the end of treatment (cycle 1 or 2; each cycle is 3 weeks) and 1 month follow-up.
  Study reports on the subjective experience of mothers with outcomes assessment visits (response to an open-question).
Change from Baseline on the feasibility of the assessment procedures - Acceptability of outcomes assessment visits (newborn-infants) | At baseline, at the end of treatment (cycle 1 or 2; each cycle is 3 weeks) and 1 month follow-up.
  Study reports on the subjective experience of mothers on the acceptability of newborn/babies acceptability of outcomes assessment visits (response to an open-question).
Estimate of recruitment | At the end of treatment (cycle 1 or 2; each cycle is 3 weeks) and 1 month follow-up.
  Study reports on recruitment
Estimate of retention | At the end of treatment (cycle 1 or 2; each cycle is 3 weeks) and 1 month follow-up.
  Study reports on retention
Estimate of dropouts | At the end of treatment (cycle 1 or 2; each cycle is 3 weeks) and 1 month follow-up.
  Study reports on dropouts
Change from Baseline in Clinical Status according to depressive symptoms. | At baseline and weekly during the 3 weeks of tDCS cycle (or during 6 weeks if tDCS cycle 2 is prescribed) and at one month follow-up
  Clinical status assessment according to Montgomery-Åsberg Depression Rating Scale (MADRS), a self report 10-item questionnaire to assess the presence and severity of clinically relevant depressive symptoms in the prior week using a 4-point scale, ranging from 0-40; higher scores mean worse clinical status
Change from Baseline in Clinical Status according to anxiety symptoms | At baseline and weekly during the 3 weeks of tDCS cycle (or during 6 weeks if tDCS cycle 2 is prescribed) and at one month follow-up
  Clinical status assessment according to Generalized Anxiety Disorder 7 (GAD-7), a 7-item tool used to screen for and assess the severity of generalized anxiety disorder in the preceding 2 weeks, rated on a 4-point scale, from 0-28 where higher scores correspond to increased presence/severity of anxiety symptoms.
Change from Baseline in Clinical Status according to difficulties in emotion regulation. | At baseline and weekly during the 3 weeks of tDCS cycle (or during 6 weeks if tDCS cycle 2 is prescribed) and at one month follow-up
  The Difficulties in Emotion Regulation Scale - Short Form (DERS) is a 18-items questionnaire to assess difficulties in using adaptive emotional regulation strategies, using a 5-point Likert scale, ranging from 18 to 72, where higher scores correspond to increased difficulties.
Change from Baseline in Clinical Status according to Sleep quality | At baseline and weekly during the 3 weeks of tDCS cycle (or during 6 weeks if tDCS cycle 2 is prescribed) and at one month follow-up
  The Pittsburgh Sleep Quality Index (PPBQ) is a 19-item questionnaire using a 4-point likert scale to assess sleep quality and disturbance over a one-month time interval, ranging between 0-57 where higher scores correspond to decreased quality of sleep.
Change from Baseline in Clinical Status according to Ruminative Thinking | At baseline and weekly during the 3 weeks of tDCS cycle (or during 6 weeks if tDCS cycle 2 is prescribed) and at one month follow-up
  The Ruminative Response Scale - Short Form7 (RRS) is a 10-item questionnaire to assess ruminative thinking, answered on a 4-point Likert scale, ranging from 0-30 where higher scores correspond to increased presence of ruminative thinking processes
Infant and Toddler Development | At baseline and 1 month follow-up
  The Bayley Scales of Infant and Toddler Development will be used to assess the developmental competences of infants from 1 to 42 months of age, consisting of 5 scales: Cognitive, Language, Motor, and Social-emotional and an Adaptive behaviour questionnaire that is completed by the mother. Composite scores are derived for cognitive, language, and motor development and scaled to a metric, with a mean of 100, standard deviation of 15, and range of 40 to 160.
Change from Baseline in bonding quality in mother-baby dyad. | At week 1, week 3 (and week 6 if two tDCS cycles where prescribed; each cycle is 3 weeks) of treatment and at 1 month follow-up.
  The Postpartum Bonding Questionnaire is a self-report 25-item questionnaire to assess early indication of disorders within mother-infant relationships, to be rated in a 5-point Likert scale. Higher scores correspond to increased dysfunction of the dyad.
Change from Baseline in parental stress. | At week 1, week 3 (and week 6 if two tDCS cycles where prescribed; each cycle is 3 weeks) of treatment and at 1 month follow-up.
  Parenting Stress Index (PSI) will be used to measure the relative stress in the parent-child relationship, primarily intended for parents of children 0-3 years. The PSI consists of a 120-item test with an optional 19-item Life Stress Scale. Its scores range between 15 and 100, and higher scores correspond to increased parental stress.
Quality of Life according to the EuroQol five dimensions, five level questionnaire - EQ-5D-5L | At baseline and 1 month follow-up
  The EQ-5D-5L is a widely used questionnaire in clinical trials, observational studies and other health surveys. The questionnaire consists of a visual analogue scale and five questions (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with five answer alternatives each. There are 3^5 = 243 combinations of the levels, each of which can be described with a five-digit number, such that the pattern 11111, indicates the optimal health state and the pattern 55555 indicates the worse health state possible.
Mother epigenetic biomarkers (collected during at-home visits) | At baseline and 1 month follow-up
  Epigenetic modifications of different neuroinflammatory genes (DNA methylation [DNAm] ) will be analysed. Saliva samples will be collected using ORAGene® (OG-500) device (for DNA extraction).
Mother genetic biomarkers (collected during at-home visits) | At baseline
  Genetic variations in the serotonin transporter gene SLC6A4 will be anlysed by sequencing analysis. Saliva samples will be collected using ORAGene® (OG-500) device (for DNA extraction).
Quantification of neuroinflammatory biomarkers of mothers (collected during at-home visits) | At baseline and 1 month follow-up
  Quantification of around 200 neuroinflammatory biomarkers will be analysed. Saliva samples will be collected using roll cotton device Salivettes (for protein analysis) and hair samples (for cortisol analysis).
Baby epigenetic biomarkers (collected during at-home visits) | At baseline and 1 month follow-up
  Epigenetic modifications of different neuroinflammatory genes (DNA methylation [DNAm] ) will be analysed. Saliva samples will be collected using ORAGene® (OG-500) device (for DNA extraction).
Quantification of neuroinflamatory biomarkers of babies (collected during at-home visits) | At baseline and 1 month follow-up
  Quantification of around 200 neuroinflammatory biomarkers will be analysed. Saliva samples will be collected using roll cotton device Salivettes (for protein analysis).
Baby genetic biomarkers (collected during at-home visits) | At baseline
  Genetic variations in the serotonin transporter gene SLC6A4 will be anlysed by sequencing analysis. Saliva samples will be collected using ORAGene® (OG-500) device (for DNA extraction).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Ganho-Ávila, PhD, Principal Investigator — University of Coimbra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] European Parliament A8-0380/2016. (2017). European Union. https://www.europarl.europa.eu/doceo /document/TA-8-2017-0028_EN.html
- [Background] Borrione L, Bellini H, Razza LB, Avila AG, Baeken C, Brem AK, Busatto G, Carvalho AF, Chekroud A, Daskalakis ZJ, Deng ZD, Downar J, Gattaz W, Loo C, Lotufo PA, Martin MDGM, McClintock SM, O'Shea J, Padberg F, Passos IC, Salum GA, Vanderhasselt MA, Fraguas R, Bensenor I, Valiengo L, Brunoni AR. Precision non-implantable neuromodulation therapies: a perspective for the depressed brain. Braz J Psychiatry. 2020 Aug;42(4):403-419. doi: 10.1590/1516-4446-2019-0741. Epub 2020 Mar 16. PMID 32187319
- [Background] Alonzo A, Fong J, Ball N, Martin D, Chand N, Loo C. Pilot trial of home-administered transcranial direct current stimulation for the treatment of depression. J Affect Disord. 2019 Jun 1;252:475-483. doi: 10.1016/j.jad.2019.04.041. Epub 2019 Apr 10. PMID 31005790
- [Background] Riggs A, Patel V, Paneri B, Portenoy RK, Bikson M, Knotkova H. At-Home Transcranial Direct Current Stimulation (tDCS) With Telehealth Support for Symptom Control in Chronically-Ill Patients With Multiple Symptoms. Front Behav Neurosci. 2018 May 22;12:93. doi: 10.3389/fnbeh.2018.00093. eCollection 2018. PMID 29872381
- [Background] Bennabi D, Haffen E. Transcranial Direct Current Stimulation (tDCS): A Promising Treatment for Major Depressive Disorder? Brain Sci. 2018 May 6;8(5):81. doi: 10.3390/brainsci8050081. PMID 29734768
- [Background] Johannsen BM, Larsen JT, Laursen TM, Bergink V, Meltzer-Brody S, Munk-Olsen T. All-Cause Mortality in Women With Severe Postpartum Psychiatric Disorders. Am J Psychiatry. 2016 Jun 1;173(6):635-42. doi: 10.1176/appi.ajp.2015.14121510. Epub 2016 Mar 4. PMID 26940804
- [Background] Molenaar NM, Kamperman AM, Boyce P, Bergink V. Guidelines on treatment of perinatal depression with antidepressants: An international review. Aust N Z J Psychiatry. 2018 Apr;52(4):320-327. doi: 10.1177/0004867418762057. Epub 2018 Mar 5. PMID 29506399
- [Background] Kim DR, Epperson CN, Weiss AR, Wisner KL. Pharmacotherapy of postpartum depression: an update. Expert Opin Pharmacother. 2014 Jun;15(9):1223-34. doi: 10.1517/14656566.2014.911842. Epub 2014 Apr 29. PMID 24773410
- [Background] Sambrook Smith M, Lawrence V, Sadler E, Easter A. Barriers to accessing mental health services for women with perinatal mental illness: systematic review and meta-synthesis of qualitative studies in the UK. BMJ Open. 2019 Jan 24;9(1):e024803. doi: 10.1136/bmjopen-2018-024803. PMID 30679296
- [Background] Wisner KL, Sit DK, McShea MC, Rizzo DM, Zoretich RA, Hughes CL, Eng HF, Luther JF, Wisniewski SR, Costantino ML, Confer AL, Moses-Kolko EL, Famy CS, Hanusa BH. Onset timing, thoughts of self-harm, and diagnoses in postpartum women with screen-positive depression findings. JAMA Psychiatry. 2013 May;70(5):490-8. doi: 10.1001/jamapsychiatry.2013.87. PMID 23487258
- [Background] Rigonatti SP, Boggio PS, Myczkowski ML, Otta E, Fiquer JT, Ribeiro RB, Nitsche MA, Pascual-Leone A, Fregni F. Transcranial direct stimulation and fluoxetine for the treatment of depression. Eur Psychiatry. 2008 Jan;23(1):74-6. doi: 10.1016/j.eurpsy.2007.09.006. Epub 2007 Nov 19. No abstract available. PMID 18023968
- [Background] Bikson M, Grossman P, Zannou AL, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Response to letter to the editor: Safety of transcranial direct current stimulation: Evidence based update 2016. Brain Stimul. 2017 Sep-Oct;10(5):986-987. doi: 10.1016/j.brs.2017.06.007. Epub 2017 Jul 12. No abstract available. PMID 28734680
- [Background] Padberg F, Kumpf U, Mansmann U, Palm U, Plewnia C, Langguth B, Zwanzger P, Fallgatter A, Nolden J, Burger M, Keeser D, Rupprecht R, Falkai P, Hasan A, Egert S, Bajbouj M. Prefrontal transcranial direct current stimulation (tDCS) as treatment for major depression: study design and methodology of a multicenter triple blind randomized placebo controlled trial (DepressionDC). Eur Arch Psychiatry Clin Neurosci. 2017 Dec;267(8):751-766. doi: 10.1007/s00406-017-0769-y. Epub 2017 Feb 28. PMID 28246891
- [Background] Cole J, Bright K, Gagnon L, McGirr A. A systematic review of the safety and effectiveness of repetitive transcranial magnetic stimulation in the treatment of peripartum depression. J Psychiatr Res. 2019 Aug;115:142-150. doi: 10.1016/j.jpsychires.2019.05.015. Epub 2019 May 16. PMID 31129438
- [Background] Garcia KS, Flynn P, Pierce KJ, Caudle M. Repetitive transcranial magnetic stimulation treats postpartum depression. Brain Stimul. 2010 Jan;3(1):36-41. doi: 10.1016/j.brs.2009.06.001. Epub 2009 Jul 8. PMID 20633429
- [Background] Vigod SN, Murphy KE, Dennis CL, Oberlander TF, Ray JG, Daskalakis ZJ, Blumberger DM. Transcranial direct current stimulation (tDCS) for depression in pregnancy: A pilot randomized controlled trial. Brain Stimul. 2019 Nov-Dec;12(6):1475-1483. doi: 10.1016/j.brs.2019.06.019. Epub 2019 Jun 19. PMID 31257092
- [Background] Sreeraj VS, Bose A, Shanbhag V, Narayanaswamy JC, Venkatasubramanian G, Benegal V. Monotherapy With tDCS for Treatment of Depressive Episode During Pregnancy: A Case Report. Brain Stimul. 2016 May-Jun;9(3):457-458. doi: 10.1016/j.brs.2016.03.007. Epub 2016 Mar 11. No abstract available. PMID 27053386
- [Background] Buchanan DM, Robaey P, D'Angiulli A. What Do We Know about Transcranial Direct Current Stimulation for Major Depression? Brain Sci. 2020 Jul 25;10(8):480. doi: 10.3390/brainsci10080480. PMID 32722399
- [Background] de Wit M, Cooper C, Reginster JY; WHO-ESCEO Working Group. Practical guidance for patient-centred health research. Lancet. 2019 Mar 16;393(10176):1095-1096. doi: 10.1016/S0140-6736(19)30034-0. Epub 2019 Mar 14. No abstract available. PMID 30894262
- [Background] Figueiredo FP, Parada AP, de Araujo LF, Silva WA Jr, Del-Ben CM. The Influence of genetic factors on peripartum depression: A systematic review. J Affect Disord. 2015 Feb 1;172:265-73. doi: 10.1016/j.jad.2014.10.016. Epub 2014 Oct 19. PMID 25451426
- [Background] Okada S, Morinobu S, Fuchikami M, Segawa M, Yokomaku K, Kataoka T, Okamoto Y, Yamawaki S, Inoue T, Kusumi I, Koyama T, Tsuchiyama K, Terao T, Kokubo Y, Mimura M. The potential of SLC6A4 gene methylation analysis for the diagnosis and treatment of major depression. J Psychiatr Res. 2014 Jun;53:47-53. doi: 10.1016/j.jpsychires.2014.02.002. Epub 2014 Feb 21. PMID 24657235
- [Background] Devlin NJ, Shah KK, Feng Y, Mulhern B, van Hout B. Valuing health-related quality of life: An EQ-5D-5L value set for England. Health Econ. 2018 Jan;27(1):7-22. doi: 10.1002/hec.3564. Epub 2017 Aug 22. PMID 28833869
- [Background] Bikson M, Hanlon CA, Woods AJ, Gillick BT, Charvet L, Lamm C, Madeo G, Holczer A, Almeida J, Antal A, Ay MR, Baeken C, Blumberger DM, Campanella S, Camprodon JA, Christiansen L, Loo C, Crinion JT, Fitzgerald P, Gallimberti L, Ghobadi-Azbari P, Ghodratitoostani I, Grabner RH, Hartwigsen G, Hirata A, Kirton A, Knotkova H, Krupitsky E, Marangolo P, Nakamura-Palacios EM, Potok W, Praharaj SK, Ruff CC, Schlaug G, Siebner HR, Stagg CJ, Thielscher A, Wenderoth N, Yuan TF, Zhang X, Ekhtiari H. Guidelines for TMS/tES clinical services and research through the COVID-19 pandemic. Brain Stimul. 2020 Jul-Aug;13(4):1124-1149. doi: 10.1016/j.brs.2020.05.010. Epub 2020 May 12. PMID 32413554
- [Background] Charvet LE, Kasschau M, Datta A, Knotkova H, Stevens MC, Alonzo A, Loo C, Krull KR, Bikson M. Remotely-supervised transcranial direct current stimulation (tDCS) for clinical trials: guidelines for technology and protocols. Front Syst Neurosci. 2015 Mar 17;9:26. doi: 10.3389/fnsys.2015.00026. eCollection 2015. PMID 25852494
- [Background] Knotkova H., Nitsche M., Bikson M., Woods A. (2019). Home-Based Patient-Delivered Remotely Supervised Transcranial Direct Current Stimulation. In Practical Guide to Transcranial Direct Current Stimulation-Principles, Procedures and Applications. Springer. https://www.springer.com/gp/book/9783319959474
- [Background] Fonseca A, Gorayeb R, Canavarro MC. Women's use of online resources and acceptance of e-mental health tools during the perinatal period. Int J Med Inform. 2016 Oct;94:228-36. doi: 10.1016/j.ijmedinf.2016.07.016. Epub 2016 Aug 3. PMID 27573331
- [Background] Tickle-Degnen L. Nuts and bolts of conducting feasibility studies. Am J Occup Ther. 2013 Mar-Apr;67(2):171-6. doi: 10.5014/ajot.2013.006270. PMID 23433271
- [Background] Orsmond GI, Cohn ES. The Distinctive Features of a Feasibility Study: Objectives and Guiding Questions. OTJR (Thorofare N J). 2015 Jul;35(3):169-77. doi: 10.1177/1539449215578649. PMID 26594739
- [Background] Seibt O, Brunoni AR, Huang Y, Bikson M. The Pursuit of DLPFC: Non-neuronavigated Methods to Target the Left Dorsolateral Pre-frontal Cortex With Symmetric Bicephalic Transcranial Direct Current Stimulation (tDCS). Brain Stimul. 2015 May-Jun;8(3):590-602. doi: 10.1016/j.brs.2015.01.401. Epub 2015 Jan 16. PMID 25862601
- [Background] Brunoni AR, Moffa AH, Sampaio-Junior B, Borrione L, Moreno ML, Fernandes RA, Veronezi BP, Nogueira BS, Aparicio LVM, Razza LB, Chamorro R, Tort LC, Fraguas R, Lotufo PA, Gattaz WF, Fregni F, Bensenor IM; ELECT-TDCS Investigators. Trial of Electrical Direct-Current Therapy versus Escitalopram for Depression. N Engl J Med. 2017 Jun 29;376(26):2523-2533. doi: 10.1056/NEJMoa1612999. PMID 28657871